CLINICAL TRIAL: NCT04339153
Title: Feasibility Study on Parents Skill Training Program for Reducing Parental Distress and Disruptive Behavior of Their Children With Autism Spectrum Disorder (ASD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2020/2
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Autism Spectrum Disorder; Disruptive Behaviours
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The study is a Randomized Controlled Trial (RCT) with single blind rating. The participants will be randomly divided into two groups. One group will receive the Parent Training (PT) and the other will get the Parent Education (PE).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Training (PT) (Experimental): The goal of intervention plan is to teach the basic applied behaviour analysis techniques to find out the antecedent of the problem behaviour, enhance adaptive skills and reduce noncompliance. Sessions will be interactive, and action-oriented through the provision of workbooks, modelling, videos, rehearsal (with child when present), homework tasks, and feedback (Bearss et al., 2015). The parents will be trained on the protocol and delivered 60 to 90 minutes preferably individual sessions over 24 weeks.
  Interventions: Behavioral: Parent Training for Disruptive Behaviours
- Parent Education (PE) (No Intervention): The Parent education group will serve as an attention-placebo condition to control for general effects of the intervention.
  There will be 12 core sessions and 1 home visit regarding knowledge of autism, learning about the principles of managing behavior, teaching new skills; improving social interaction and communication. Each session will last for 60 to 90 minutes over 24 weeks.

INTERVENTIONS:
Behavioral: Parent Training for Disruptive Behaviours — Critically, PT also involves education about autism during the initial sessions, and thus benefits of PT are inferred to come from the specific training.
  Arms: Parent Training (PT)

SUMMARY:
Children with Autism Spectrum Disorder (ASD) usually exhibt problematic behavioral issues such as hitting, non-compliance, tantrums, spitting, headbanging and aggression, this not only cause distress for the child but also has a significant effect on the mental health of the parents.

In Pakistan, the rise in ASD children, lack of resources, non-advocacy, and limited knowledge amongst health professionals have created an alarming situation not only psychologically but also because of the economic burden. The current study is to assess the impact of a psychoeducation and parental skills training programme for reducing the parental psychological stress and disruptive behavior of their children with Autism. This is a 24 weeks parent education and behavioural management manualized programme based on the principles of applied behavior analysis.

The plan will include skills training on replacing problematic behaviours with more appropriate behaviours, improving social communication in verbal and non-verbal children, and interactions with peers and others. The parents will be trained on the manualized training programme in groups or as individual sessions using modelling, role-plays and rehearsal as training methods. A total of 60 parents of ASD children, age ranges from 3 to 9 years with disruptive behaviour will be recruited. The diagnosed ASD children screened from the standardised instruments not later than six months and scored > 15 on the subscale Irritability of Aberrant Behaviour Checklist will be randomly divided into two groups, 1) parents receiving manualized training program 2) parents receiving education sessions. The baseline will be determined baseline by using parent-rated instruments for behavioural problems using the Aberrant Behaviour Checklist, Home Situation Questionnaire, Vineland Adaptive behaviour scales, Symptom Checklist 90, and Parental Distress Index. Overall there will be 12 core sessions on the Parental Education (PE) pertaining to parent education including advocacy and educational planning over 24 weeks and 11 sessions of Parent Training (PT) for managing behavioural issues of autistic children. Each session will last for 60 to 90 minutes. There will be six months follow up, and evaluation will be done by the masked assessor. All the sessions will be from a trained psychologist and behaviour analysts who have more than 1 year experience of working with children with ASD. To ensure treatment integrity, all training sessions will be assessed after every 4 weeks by using behavioural measures to evaluate the correct implementation of treatment protocol. Some of the sessions will be recorded.

It is anticipated that parent training will improve the mental health of parents and reduce the disruptive behaviour of children with Autism Spectrum Disorder.

ELIGIBILITY:
Inclusion Criteria:

Children aged 3 to 9 years will be recruited. The gold standard diagnostic tools i.e. the autism diagnostic observation schedule (ADOS) will be administered by a trained assessor to confirm the diagnosis of ASD.

To ensure our intervention reaches children with behavioural difficulties, children who will score > 15 on the subscale of Irritability ABC-C will be included.

Exclusion Criteria:

Potential participants with an intellectual disability and non-receptive, or who have a severe medical illness will be excluded from the study.

Although unlikely to occur, children with ASD whose parents have received any intensive parent training during the past 24 months will not be included

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-04-02 (Estimated); Primary Completion 2021-09-02 (Estimated); Study Completion 2021-09-02 (Estimated)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist-Community (ABC-C; Aman & Singh, 1994) | 24 weeks
  The ABC is an informant scale rated 0 to 3 for assessing problem behaviour scales. Its subscales and respective numbers of items are as follows: 1. Irritability (15 items), 2. Social Withdrawal (16 items), 3. Stereotypic Behavior (7 items), 4. Hyperactivity/Noncompliance (16 items), and 5. Repetitive Speech (4 items).
Parenting Stress Index, Fourth Edition Short Form (PSI-4; Abidin, 1995) | 24 weeks
  It is a 120-item measure used to examine parental stress levels considering a parent's relationship with one of his or her children between the ages of 1 month and 12 years. There are three domains i.e, (a) child characteristics, (b) parent characteristics, and (c) situational/demographic life stress.
Symptom Checklist-90 (SCL-90, Derogatis, Rickels, Rock, 1976) | 24 weeks
  The SCL-90 will be used to measure the psychological distress. It is also a valid measure of screening nine symptoms including somatization, hostility, depression, anxiety, interpersonal sensitivity, social anxiety, paranoia, obsessive compulsive and agoraphobia. Sum of all the subscales indicate the psychological distress and having .98 reliability which is highly satisfactory.

SECONDARY OUTCOMES:
Vineland Adaptive Behavior Scales (Vineland-II; Sparrow, Cicchetti, & Balla, 2005) | 24 weeks
  It is used to evaluate the four broad domains including communication, daily living skills, socialization and motor skills. It also includes an optional scale to assess maladaptive behaviour.
Home Situations Questionnaire Disorder (HSQ; Chowdhury et al, 2016) | 24 weeks
  It is a 24-item parent rating scale from 1 (mild) to 9 (severe). It is designed to evaluate noncompliance in children with ASD.
Clinical Global Impressions - Improvement Scale (CGI; Guy 1976) | 24 weeks
  It is a 7-point scale designed to measure overall improvement from baseline. Scores range from 1 (very much improved) through 4 (unchanged) to 7 (very much worse). Scores of 1 or 2 at week 24 endpoint identified clinical responders.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Shafique, Dr, Principal Investigator — FUI; Nasim Chaudhary, Dr. Prof., Study Chair — FUI; Nusrat Hussain, Dr. Prof., Principal Investigator — University of Manchester; Jumana Ahmad, Principal Investigator — Greenwich University

IPD SHARING:
Plan to Share IPD: No